CLINICAL TRIAL: NCT02425904
Title: Phase II Study of Clofarabine in Patients With Recurrent or Refractory Langerhans Cell Histiocytosis and LCH-related Disorders
Brief Title: Study of Clofarabine in Patients With Recurrent or Refractory Langerhans Cell Histiocytosis and LCH-related Disorders
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Sanofi (Industry); St. Baldrick's Foundation (Other); Cookies for Kids' Cancer (Other); North American Consortium for Histiocytosis (Other)
Responsible Party: Principal Investigator, Barbara Degar, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-005
Record Dates: First submitted 2015-04-18; First posted 2015-04-24 (Estimated); Results first posted 2022-02-16 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: Langerhans Cell Histiocytosis
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recurrent or Refractory Langerhans Cell Histiocytosis (LCH) + Clofarabine (Experimental): Participants with recurrent or refractory LCH defined as with multi-focal or multi-system disease who have recurred (or have refractory disease) after at least one prior systemic chemotherapy regimen.
  Patient will receive Clofarabine administered via IV on days 1-5, 25 mg/m2/day per cycle for 2 cycles. At the end of cycle 2 if no disease progression, will continue with same dose for maintenance treatment for 4 additional cycles.
  Interventions: Drug: Clofarabine
- LCH-related disorders + Clofarabine (Experimental): Participants with LCH-related disorders defined as who require systemic chemotherapy including participants with Rosai Dorfman Disease (RDD) who have not responded to or recurred after treatment with corticosteroids. Erdheim Chester Disease (ECD) subjects who have confirmed presence of BRAF V600E mutation must have not responded to, have recurred after, or be unable to receive treatment with a BRAF inhibitor.
  Patient will receive Clofarabine administered via IV on days 1-5, 25 mg/m2/day per cycle for 2 cycles. At the end of cycle 2 if no disease progression, will continue with same dose for maintenance treatment for 4 additional cycles.
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — second-generation purine nucleoside analog
  Other Names: Clofarex; Clolar

SUMMARY:
This research study is evaluating a drug called clofarabine as a possible treatment for Langerhans Cell Histiocytosis (LCH) and and other histiocytic disorders.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational intervention, to learn whether the drug works in treating a specific disease, in this case, clofarabine to treat LCH.

"Investigational" means that the intervention is still being studied. It also means that the FDA (the U.S. Food and Drug Administration) has not yet approved clofarabine for your disease.

Clofarabine is a chemotherapy drug that has been used and is approved by the FDA for the treatment of leukemia in children and adults. Information from other research studies suggests that this drug may also be effective in participants with LCH and other histiocytic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of Langerhans Cell Histiocytosis (stratum 1) or LCH-related disorder (stratum 2) established by standard diagnostic criteria and confirmed histologically.
* Evidence of active disease (histological confirmation of reactivation or progression is not required).
* Performance Score > 70% (use Lansky score for age < 16 and Karnofsky score for age = >16).
* Patients of all ages will be eligible.
* Provide signed written informed consent.
* In stratum 1, patients must have failed one prior systemic chemotherapy regimen. In stratum 2, RDD patients must have failed treatment with corticosteroid. ECD patients who have confirmed BRAF V600E mutation must have failed treatment with a BRAF inhibitor or are not considered to be eligible for such treatment.
* There is no limitation of amount or the type of prior therapy or drugs.
* Female patients of childbearing potential must have a negative serum pregnancy test within 14 days prior to enrollment. Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
* Participants must have adequate marrow functions as defined below, except those with involvement of hematopoietic system for whom these criteria can be waived:

  * Absolute neutrophil count ≥ 750 cells/µL
  * Platelets ≥75,000/µL
* Participants must have adequate organ functions as defined below:

  * Total bilirubin ≤ 2.5x institutional upper limit of normal
  * AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal unless it is related to involvement by LCH
  * Adequate renal function defined as:
  * Pediatric Population (patients < 18 years): Creatinine within normal limits or calculated creatinine clearance greater than or equal to 90 ml/min/1.73 m2 as calculated by the Schwartz formula for estimated glomerular filtration rate (GFR) where GFR (ml/min/1.73 m2) = k x Height (cm)/serum creatinine (mg/dl). k is a proportionality constant which varies with age and is a function of urinary creatinine excretion per unit of body size; 0.45 up to 12 months of age; 0.55 children and adolescent girls; and 0.70 adolescent boys.
  * Adult Population (patients >= 18 years): Serum creatinine less than or equal to 1.0 mg/dL; if serum creatinine >1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be >60 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation where Predicted GFR (ml/min/1.73 m2) = 186 x (Serum Creatinine)-1.154 x (age in years)-0.203 x (0.742 if patient is female) x (1.212 if patient is black), where serum creatinine is measured in mg/dL.
  * Alkaline phosphatase ≤ 2.5 x institutional upper limit of normal

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier. Corticosteroid treatment is allowed.
* Participants may not be receiving any other investigational agents targeting Histiocytosis.
* Clofarabine is excreted primarily by the kidneys. Therefore, drugs with known renal toxicity (e.g.vancomycin, amphotericin B, acyclovir, cyclosporin, methotrexate, tacrolimus) should be avoided to the extent possible during the 5 days of clofarabine treatment in each cycle or, if required, administered cautiously and with close monitoring.
* Use of alternative medications (e.g., herbal or botanical that could interfere with clofarabine) is not permitted during the entire study period.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because clofarabine is a nucleoside analog with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with clofarabine, breastfeeding should be discontinued if the mother is treated with clofarabine. These potential risks may also apply to other agents used in this study.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Patients with a history of prior hematopoietic stem cell transplantation (HSCT), elevated conjugated serum bilirubin at study entry, uncontrolled systemic fungal, bacterial, or other infection, a history of hepatitis B or C infection or a history of cirrhosis.
* Individuals who are known to be HIV-positive on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with clofarabine. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Degar, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (14):
- United States (13):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mount Sinai Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
- The Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: from 5/21/2015 to 1/14/2020
Period: Overall Study
Arm/Group | Recurrent or Refractory Langerhans Cell Histiocytosis (LCH) + Clofarabine | LCH-related Disorders + Clofarabine
Started | 20 | 5
Efficacy Analysis | 20 | 4 (1 patient was incorrectly assigned to LCH-related disorders cohort but it is actually LCH patients, so excluded from efficacy analysis.)
Completed | 17 | 2
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recurrent or Refractory Langerhans Cell Histiocytosis (LCH) + Clofarabine | LCH-related Disorders + Clofarabine | Total
Number analyzed (Participants) | 20 | 5 | 25
Age, Customized [Median (Full Range); unit: years] | 3.4 [0.6 to 10.6] | 38.6 [10.7 to 58.2] | 4.3 [0.6 to 58.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 2 | 17
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 15 | 5 | 20
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 17 | 5 | 22
  Canada | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (OR) of LCH Cohort
Description: The OR was defined as the proportion of participants achieving certain response on treatment among LCH patients, criteria were defined per protocol. Better response were defined as achieving complete disease resolution (NAD) or disease regression (AD better); intermediate response defined as stable or unchanged disease status; worse response defined as disease progression.
Time Frame: Disease was evaluated at baseline and the end of cycle 2. Treatment continued after cycle 2 until disease progression or unacceptable toxicity. LCH treatment duration has a median of 5.8 months with range 2.1-7 months.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Recurrent or Refractory Langerhans Cell Histiocytosis (LCH) + Clofarabine
Number analyzed (Participants) | 20
proportion of participants
  Better | 0.85 [0.62 to 0.97]
  Intermediate | 0.15 [0.03 to 0.38]
  Worse | 0 [0 to 0]

2. Primary Outcome: Response Rate of LCH-related Disorders Cohort
Description: The OR was defined as the proportion of participants achieving certain response on treatment among LCH-related disorder patients, criteria were defined per protocol. A clinical response of progressive metabolic disease (PMD) defined as CT-based target lesion abnormal and bone marrow new or recurrent involvement; partial metabolic response (PMR) defined as CT-based target lesion decreasing or disease regressed.
Time Frame: Disease was evaluated at baseline and the end of cycle 2. Treatment continued after cycle 2 until disease progression or unacceptable toxicity. Treatment duration has a median of 5.5 months with range 1.7-5.6 months.
Population: 1 patient excluded because of problematic enrollment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | LCH-related Disorders + Clofarabine
Number analyzed (Participants) | 4
proportion of participants
  PMR | 0.75 [0.19 to 0.99]
  PMD | 0.26 [0.006 to 0.81]

3. Secondary Outcome: 1-year Progression Free Survival (PFS)
Description: 1-year PFS defined as the proportion of patients that survival progression free at 1 year. PFS based on the duration of time from study entry to documented disease progression (PD) or death. Per protocol criteria: where time to event for PFS is the time from study enrollment until the time of first occurrence of new lesions, progressive disease, or death from any cause, or until last contact if no event occurs.
Time Frame: At 1 year
Measure: Number; unit: proportion of patients
Arm/Group | Recurrent or Refractory Langerhans Cell Histiocytosis (LCH) + Clofarabine | LCH-related Disorders + Clofarabine
Number analyzed (Participants) | 20 | 4
proportion of patients | 0.89 | 0.5

4. Secondary Outcome: 1-year Overall Survival (OS)
Description: 1-year OS defined as the proportion of patients that survival at 1 year. OS calculated as the time from enrollment until death or censored at date last known alive.
Time Frame: At 1 year
Measure: Number; unit: proportion of patients
Arm/Group | Recurrent or Refractory Langerhans Cell Histiocytosis (LCH) + Clofarabine | LCH-related Disorders + Clofarabine
Number analyzed (Participants) | 20 | 4
proportion of patients | 1 | 0.75

5. Secondary Outcome: Number of Participants With at Least One Grade 3 or Higher Treatment-Related Toxicity
Description: All grade 3 or higher adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4.0 as reported on case report forms were counted. Number of Participants with at least one Grade 3 or Higher Treatment-Related Toxicity defined as number of patients experiencing at least one treatment-related grade 3 or higher AE of any type during the time of observation.
Time Frame: Disease was evaluated at baseline and the end of cycle 2. Treatment continued after cycle 2 until disease progression or unacceptable toxicity. LCH treatment duration is median 5.8 with range 2.1-7 months; LCH-related treatment duration is 5.5 (1.7-5.6).
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent or Refractory Langerhans Cell Histiocytosis (LCH) + Clofarabine | LCH-related Disorders + Clofarabine
Number analyzed (Participants) | 20 | 4
Participants | 15 | 4

ADVERSE EVENTS:
Time Frame: Adverse events are assessed every cycle until the end of treatment. LCH Cohort treatment duration has a median of 5.8 months with range 2.1-7 months. LCH-related Disorders Cohort Treatment duration has a median of 5.5 months with range 1.7-5.6 months.
Description: Serious adverse events (AEs) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Maximum grade toxicity by type for a patient over time was calculated. No further data is available to specify classification of other beyond the general term.
Groups:
- Recurrent or Refractory Langerhans Cell Histiocytosis (LCH) + Clofarabine: Participants with recurrent or refractory LCH defined as with multi-focal or multi-system disease who have recurred (or have refractory disease) after at least one prior systemic chemotherapy regimen.
  Patient will receive Clofarabine administered via IV on days 1-5, 25 mg/m2/day per cycle for 2 cycles. At the end of cycle 2 if no disease progression, will continue with same dose for maintenance treatment for 4 additional cycles.
  Clofarabine: second-generation purine nucleoside analog
- LCH-related Disorders + Clofarabine: Participants with LCH-related disorders defined as who require systemic chemotherapy including participants with Rosai Dorfman Disease (RDD) who have not responded to or recurred after treatment with corticosteroids. Erdheim Chester Disease (ECD) subjects who have confirmed presence of BRAF V600E mutation must have not responded to, have recurred after, or be unable to receive treatment with a BRAF inhibitor.
  Patient will receive Clofarabine administered via IV on days 1-5, 25 mg/m2/day per cycle for 2 cycles. At the end of cycle 2 if no disease progression, will continue with same dose for maintenance treatment for 4 additional cycles.
  Clofarabine: second-generation purine nucleoside analog
Arm/Group | Recurrent or Refractory Langerhans Cell Histiocytosis (LCH) + Clofarabine | LCH-related Disorders + Clofarabine
All-Cause Mortality (participants affected / at risk) | 0/20 | 3/4
Serious Adverse Events (participants affected / at risk) | 15/20 | 4/4
Other Adverse Events (participants affected / at risk) | 20/20 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Recurrent or Refractory Langerhans Cell Histiocytosis (LCH) + Clofarabine (N=20) | LCH-related Disorders + Clofarabine (N=4)
Alanine aminotransferase increased (Investigations) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 8 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 0/0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0/0
Hyponatremia (Metabolism and nutrition disorders) | 0/0 | 1
Lung infection (Infections and infestations) | 0/0 | 1
Lymphocyte count decreased (Investigations) | 3 | 1
Mucosal infection (Infections and infestations) | 1 | 0/0
Mucositis oral (Gastrointestinal disorders) | 1 | 0/0
Neutrophil count decreased (Investigations) | 8 | 2
Oral pain (Gastrointestinal disorders) | 1 | 0/0
Platelet count decreased (Investigations) | 3 | 4
Urinary tract infection (Infections and infestations) | 1 | 0/0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0/0
Vomiting (Gastrointestinal disorders) | 1 | 0/0
White blood cell decreased (Investigations) | 4 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Recurrent or Refractory Langerhans Cell Histiocytosis (LCH) + Clofarabine (N=20) | LCH-related Disorders + Clofarabine (N=4)
Abdominal distension (Gastrointestinal disorders) | 1 | 0/0
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Agitation (Psychiatric disorders) | 1 | 0/0
Alanine aminotransferase increased (Investigations) | 0/0 | 1
Alkaline phosphatase increased (Investigations) | 0/0 | 1
Allergic reaction (Immune system disorders) | 2 | 0/0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0/0
Anal pain (Gastrointestinal disorders) | 1 | 0/0
Anemia (Blood and lymphatic system disorders) | 5 | 2
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0/0
Aspartate aminotransferase increased (Investigations) | 1 | 2
Ataxia (Nervous system disorders) | 1 | 0/0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0/0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0/0
Confusion (Psychiatric disorders) | 0/0 | 1
Conjunctivitis (Eye disorders) | 1 | 0/0
Constipation (Gastrointestinal disorders) | 11 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 0/0
Creatinine increased (Investigations) | 1 | 0/0
Dental caries (Gastrointestinal disorders) | 1 | 0/0
Depression (Psychiatric disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 7 | 0/0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0/0
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0/0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 2 | 0/0
Ear pain (Ear and labyrinth disorders) | 4 | 0/0
Edema face (General disorders) | 0/0 | 1
Edema limbs (General disorders) | 1 | 0/0
Edema trunk (General disorders) | 1 | 0/0
Endocrine disorders - Other, specify (Endocrine disorders) | 3 | 0/0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Eye disorders - Other, specify (Eye disorders) | 1 | 0/0
Eye infection (Infections and infestations) | 1 | 0/0
Fatigue (General disorders) | 9 | 3
Fever (General disorders) | 10 | 2
Flu like symptoms (General disorders) | 2 | 0/0
Gait disturbance (General disorders) | 1 | 0/0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 0/0
Headache (Nervous system disorders) | 4 | 1
Hearing impaired (Ear and labyrinth disorders) | 2 | 0/0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0/0 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0/0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0/0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0/0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0/0
Hypotension (Vascular disorders) | 2 | 0/0
Hypothyroidism (Endocrine disorders) | 0/0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0/0
Irritability (General disorders) | 2 | 0/0
Lip infection (Infections and infestations) | 1 | 0/0
Lip pain (Gastrointestinal disorders) | 1 | 0/0
Localized edema (General disorders) | 0/0 | 1
Lymphocyte count decreased (Investigations) | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0/0
Nausea (Gastrointestinal disorders) | 11 | 3
Neuralgia (Nervous system disorders) | 1 | 0/0
Neutrophil count decreased (Investigations) | 2 | 0/0
Obesity (Metabolism and nutrition disorders) | 1 | 0/0
Otitis media (Infections and infestations) | 2 | 0/0
Pain (General disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Palpitations (Cardiac disorders) | 0/0 | 1
Platelet count decreased (Investigations) | 3 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0/0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0/0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0/0
Rectal pain (Gastrointestinal disorders) | 1 | 0/0
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 0/0
Scleral disorder (Eye disorders) | 1 | 0/0
Sinus tachycardia (Cardiac disorders) | 7 | 0/0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0/0
Thromboembolic event (Vascular disorders) | 1 | 0/0
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0/0
Tremor (Nervous system disorders) | 1 | 0/0
Upper respiratory infection (Infections and infestations) | 1 | 0/0
Urinary incontinence (Renal and urinary disorders) | 1 | 0/0
Urinary tract pain (Renal and urinary disorders) | 1 | 0/0
Vaginal pain (Reproductive system and breast disorders) | 1 | 0/0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0/0 | 1
Vomiting (Gastrointestinal disorders) | 12 | 2
Weight gain (Investigations) | 1 | 0/0
Weight loss (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT02425904/Prot_SAP_000.pdf